CLINICAL TRIAL: NCT04593381
Title: Efficacy and Safety of Stereotactic Body Radiotherapy (SBRT in Oligo-metastatic/Persistent/Recurrent Ovarian Cancer (MPR-OC): a Prospective, Multicenter Phase II Study (MITO-RT3/RAD)
Brief Title: Efficacy and Safety of SBRT in Oligo-metastatic/Persistent/Recurrent Ovarian Cancer
Acronym: MITO-RT3/RAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gemelli Molise Hospital (Other)
Collaborators: Fondazione Policlinico Universitario A. Gemelli, IRCCS (Unknown)
Responsible Party: Principal Investigator, Gabriella Macchia, Radiation Oncologist, Gemelli Molise Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE 07-14-2020
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Ovarian Neoplasms; Recurrent Ovarian Carcinoma; Oligometastatic Disease
Keywords: Oligometastasis; Stereotactic body radiotherapy; SBRT; SABR
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT treatment (Experimental): Intervention: Radiation: SBRT
  Interventions: Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — All patients accrued will be treated with SBRT to all sites of active metastatic disease as per CT scan or PET/CT and/or MRI. A range of schedules and doses are provided, it is advised that the maximum dose that can be achieved whilst meeting the organs at risk planning constraints is prescribed.

SUMMARY:
This is a prospective, multicenter, Phase II study aimed at defining the activity and safety of SBRT in MPR-OC. Clinical and imaging data as well as SBRT parameters would be analyzed with the aim to identify potential predictors of response to treatment and clinical outcome.

DETAILED DESCRIPTION:
Stereotactic Body Radiotherapy (SBRT) represents the cutting edge within high conformal and modulated radiotherapy techniques; it can provide high local control (LC) for curative-intent of low burden metastatic, persistent and metastatic lesions in face of minimal acute and late toxicities. SBRT is amenable even in patients who had already been managed by radiotherapy. In addition, SBRT has been shown to be active in chemoresistant disease, and potentially able to mount immune response through the release of tumor neoantigens after cell killing, thus allowing to synergize with immunotherapeutic approaches. SBRT has been widely adopted in the clinical setting of oligometastatic/persistent/recurrent (MPR) disease (up to <5 lesions) in several malignancies including also ovarian cancer (OC); the recently published retrospective, multicenter Italian study (MITO-RT1) has confirmed the activity and safety of SBRT in MPR OC, thus providing a model able to predict the higher chance of complete response of tumor lesions to SBRT, and local control rate.

The MITO-RT3/RAD trial is a prospective, Italian multicenter Phase II study aimed at evaluating the activity and safety of SBRT in MPR-OC patients. Clinical and imaging data, as well as SBRT technical parameters, would be analyzed with the aim to identify potential predictors of response to treatment and clinical outcome: in this context, additional insights into the tissue features of tumor lesions would be of clinical interest in the context of the personalized treatment, as testified by studies demonstrating that image-based quantitative features from pre-treatment imaging could predict clinical outcomes in several malignancies.

Furthermore, given the crucial role played by the mutational status of BRCA 1/2 genes in this disease, the assessment of BRCA gene status was considered mandatory, thus representing inclusion criteria.

The study will include patients with oligo-metastatic/persistent/recurrent lesions (MPR) from OC patients for which salvage surgery or other local therapies resulted not feasible, as per relative contraindication to further systemic therapy because of serious comorbidities, as per previous severe toxicity, unavailability of potentially active chemotherapy, or patient refusal of systemic therapy

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ovarian cancer
* age >18 yrs,
* ECOG performance status 0-3,
* expected life expectancy >6 months,
* 1-5 synchronous lesions
* any site of disease,
* compulsory assessment of mutational status of BRCA1/2 genes (either germline or somatic),
* salvage surgery or other local therapies not feasible,
* relative contraindication to further systemic therapy because of serious comorbidities,
* previous severe systemic therapy toxicity
* unavailability of potentially active systemic therapy,
* patient refusal of systemic therapy,
* Re-treatment of lesions already treated with conventional external beam radiotherapy is allowed*

Exclusion Criteria:

* mucinous OC,
* borderline ovarian tumors,
* non-epithelial OC,
* previous radiotherapy severe toxicity
* co-morbidities and functional impairment considered clinically precluding the safe use of SBRT,
* pregnancy
* any psychological, sociological, or geographical issue potentially hampering compliance with the study,
* lesion diameter larger than 5 centimeters

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 376 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical complete response to SBRT by imaging | Assessment of Clinical complete response at six months
  Radiologic response will be evaluated by morphological (contrast-enhanced CT scan and/or MRI) or functional imaging modalities (18F-fluorodeoxyglucose-PET) and classified according to the RECIST (version 1.1) or PERCIST criteria.

SECONDARY OUTCOMES:
2-yr actuarial LC rate | 2 years
  progression of disease inside SBRT field on a per lesion basis
2-yr progression-free survival | 2 years
  progression of disease out of SBRT field
2-yr overall survival | 2 years
  patient survival
treatment free interval | 2 years
  time without any new treatment start after SBRT
rate of toxicity | 2 years
  SBRT acute and late toxicity rate
2-yr actuarial late toxicity free survival | 2 years
  actuarial evaluation of late toxicity

OTHER OUTCOMES:
Radiomic clusters analysis | 2 years
  Investigation of radiomic features for clustering analysis to predict response according to other histological and clinical parameters
Breast cancer genes 1/2 (BRCA genes) characterization | 2 years
  Investigation of the mutational status of BRCA 1/2 genes in this disease

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Macchia, Principal Investigator — Radiotherapy Unit, Gemelli Molise
Locations (14):
- Italy (14):
  - Responsible Research Hospital, Campobasso, CB
  - S.C. di Radioterapia Oncologica-Azienda Sanitaria locale, Biella
  - Azienda Ospedaliera "Cannizzaro", Catania
  - Azienda sanitaria locale Lanciano Vasto Chieti, Chieti
  - Ospedale Vito Fazzi, Lecce
  - Department of Radiation Oncology, IRCCS San Raffaele Scientific Institute, Milan
  - Humanitas Clinical and Research Center-IRCCS, Milan
  - Azienda USL - IRCCS di Reggio Emilia, Reggio Emilia
  - Campus Biomedico, Roma
  - Policlinico A. Gemelli, IRCCS, Roma
  - Università La Sapienza, Roma
  - Fatebenefratelli Isola Tiberina-Gemelli Isola,, Roma
  - S Maria Hospital, Terni
  - Azienda Sanitaria Universitaria Friuli Centrale (ASU FC) - SOC Radioterapia, Udine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macchia G, Lazzari R, Colombo N, Laliscia C, Capelli G, D'Agostino GR, Deodato F, Maranzano E, Ippolito E, Ronchi S, Paiar F, Scorsetti M, Cilla S, Ingargiola R, Huscher A, Cerrotta AM, Fodor A, Vicenzi L, Russo D, Borghesi S, Perrucci E, Pignata S, Aristei C, Morganti AG, Scambia G, Valentini V, Jereczek-Fossa BA, Ferrandina G. A Large, Multicenter, Retrospective Study on Efficacy and Safety of Stereotactic Body Radiotherapy (SBRT) in Oligometastatic Ovarian Cancer (MITO RT1 Study): A Collaboration of MITO, AIRO GYN, and MaNGO Groups. Oncologist. 2020 Feb;25(2):e311-e320. doi: 10.1634/theoncologist.2019-0309. Epub 2019 Oct 10. PMID 32043791
- [Derived] Macchia G, Pezzulla D, Campitelli M, Lucci S, Draghini L, Russo D, Fodor A, D'Agostino GR, Balcet V, Tamburo M, Giaccherini L, Tortoreto F, Augurio A, Ippolito E, Stefano AD, Fanelli M, Petrella L, Cilla S, Cosentino F, Marchetti C, Salutari V, Morganti AG, Gambacorta MA, Fagotti A, Pignata S, Scambia G, Ferrandina G, Deodato F. Treatment of Oligometastatic Parenchymal Lesions in Ovarian Cancer With Stereotactic Ablative Radiation Therapy: A Multicenter Prospective Phase 2 Trial (MITO RT3/RAD). Int J Radiat Oncol Biol Phys. 2025 Sep 1;123(1):228-237. doi: 10.1016/j.ijrobp.2025.03.032. Epub 2025 Mar 31. PMID 40174649
- [Derived] Macchia G, Jereczek-Fossa BA, Lazzari R, Cerrotta A, Deodato F, Ippolito E, Aristei C, Gambacorta MA, Scambia G, Valentini V, Ferrandina G. Efficacy and safety of stereotactic body radiotherapy (SBRT) in oligometastatic/persistent/recurrent ovarian cancer: a prospective, multicenter phase II study (MITO-RT3/RAD). Int J Gynecol Cancer. 2022 Jul 4;32(7):939-943. doi: 10.1136/ijgc-2021-002709. PMID 34155084